CLINICAL TRIAL: NCT05393063
Title: A Phase I Open-label Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of AK127 Monotherapy in Patients With Advanced Malignant Tumors
Brief Title: A Study to Evaluate the Efficacy and Safety of AK127 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK127-102
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK127 (Experimental): Subjects will receive AK127 by intravenous administration
  Interventions: Drug: AK127

INTERVENTIONS:
Drug: AK127 — Subjects will receive AK127 by intravenous administration（administered on Day 1 of each cycle, Q3W）
  Other Names: Subjects will receive AK127 by intravenous administration

SUMMARY:
This study is to characterize the safety, tolerability and anti-tumor activity of AK127 as a single agent in adult subjects with advanced solid tumor malignancies.

DETAILED DESCRIPTION:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of AK127 as a single agent in adult subjects with advanced solid tumor malignancies. The study, as a dose escalation phase is to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for AK127 as a single agent, and describe Dose Limiting Toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
4. Life expectancy ≥3 months.
5. Histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject is not suitable for standard therapy.
6. Adequate organ function.
7. Patients of childbearing potential must agree to use effective contraceptive measures.

Exclusion Criteria:

1. The patient has received prior immunotherapy against TIGIT target.
2. Not currently enrolled in any other clinical study.
3. Receipt of any anticancer therapy within 4 weeks or within 5 half-lives of the drug prior to the first dose of AK127.
4. Symptomatic central nervous system metastases.
5. Active malignancies within the past 1 years, with the exception of tumors in this study and cured local tumors.
6. Active autoimmune disease requiring systemic treatment prior to the start of study treatment.
7. There is a history of major diseases 1 year prior to the first dose.
8. Medical history of gastrointestinal perforation or gastrointestinal fistula within 6 months prior to the first dose.
9. Received chest radiation therapy prior to the first dose.
10. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage.
11. Active or previously documented inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
12. Receipt of live or attenuated vaccination within 4 weeks prior to the first dose of AK127.
13. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
14. Known history of active tuberculosis.
15. History of organ transplant or hematopoietic stem cell.
16. History of primary immunodeficiency.
17. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
18. Other cases deemed inappropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 21 days
  DLTs will be assessed during the first 21 days of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected or definite relationship to study drug

SECONDARY OUTCOMES:
PFS | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by investigator Per RECIST 1.1.
ORR | Up to 2 years
  Efficacy measures such as overall response rate (ORR), which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1
DCR | Up to 2 years
  Disease control rate (DCR), which is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
DOR | Up to 2 years
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
TTR | Up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
Area under the Concentration-Time Curve (AUC) of AK127 | Cycle 1 and 4: Predose, Post-dose-5min,2 hours, 24 hours, Day 4,8 and 15; Cycle 2,3,5,6: Predose and Post-dose-5min; then Predose at Day 1, every 2 cycles (cycle length 21 days),Day30 after last dose; Up to 2 years and 1 months
  The endpoints for assessment of PK of AK127 include serum concentrations of AK127 at different timepoints after AK127 administration
Maximum observed concentration (Cmax) of AK127 | Cycle 1 and 4: Predose, Post-dose-5min,2 hours, 24 hours, Day 4,8 and 15; Cycle 2,3,5,6: Predose and Post-dose-5min; then Predose at Day 1, every 2 cycles (cycle length 21 days),Day30 after last dose; Up to 2 years and 1 months
  The endpoints for assessment of PK of AK127 include serum concentrations of AK127 at different timepoints after AK127 administration
Minimum observed concentration (Cmin) of AK127 at steady state | Cycle 1 and 4: Predose, Post-dose-5min,2 hours, 24 hours, Day 4,8 and 15; Cycle 2,3,5,6: Predose and Post-dose-5min; then Predose at Day 1, every 2 cycles (cycle length 21 days),Day30 after last dose; Up to 2 years and 1 months
  The endpoints for assessment of PK of AK127 include serum concentrations of AK127 at different timepoints after AK127 administration
Number and Percentage of Subjects with Anti-Drug Antibodies(ADAs) to AK127 | Predose on Day 1 at Cycle 1-6, then Predose at Day 1, every 2 cycles,Day30 after last dose; Up to 2 years and 1 months
  The immunogenicity of AK127 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Chief doctor, Principal Investigator — Shanghai Chest Hospital; Yun Fan, Chief doctor, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No